CLINICAL TRIAL: NCT04720261
Title: Efficacy of a Personalized Caplacizumab Regimen Based on ADAMTS13 Activity Monitoring in Adult Acquired Thrombotic Thrombocytopenic Purpura: A Phase II, Multicenter Non-inferiority Single-arm Study.
Brief Title: Efficacy of a Personalized Caplacizumab Regimen Based on ADAMTS13 Activity Monitoring in Adult aTTP
Acronym: CAPLAVIE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019/0408/HP
Record Dates: First submitted 2021-01-12; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Thrombotic Thrombocytopenic Purpura, Acquired
MeSH Terms: conditions — Thrombotic thrombocytopenic purpura, acquired | interventions — caplacizumab

STUDY DESIGN:
Intervention Model Description: Experimental, prospective, non-comparative, multicentric national study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Caplacizumab (Other): All patients in the study are aTTP and needs to be treated by caplacizumab. The duration of this treatment will be evaluated through the ADAMTS 13 activity.
  Interventions: Drug: Caplacizumab

INTERVENTIONS:
Drug: Caplacizumab — Analyse of ADAMTS13 activity in patients with aTTP treated with Caplacizumab in order to help adapting the treatment with caplacizumab in TTP patients

SUMMARY:
The aim of the study is to evaluate the efficacy of a personalized caplacizumab regimen based on ADAMTS13 activity monitoring in adult acquired thrombotic thrombocytopenic purpura (aTTP): This study is a phase II, prospective, multicenter non-inferiority single-arm study.

DETAILED DESCRIPTION:
ADAMTS13 activity will be evaluated on day 7 after the end of daily PE and every 7 days until ADAMTS13 activity ≥ 20% is reached. In case of persistent severe ADAMTS13 deficiency (≤ 20%), caplacizumab administration could be extended for a maximum of 58 days after the end of the daily PE period and should be accompanied by an adjusted immunosuppressive therapy as needed. This duration is in accordance with the HERCULES study protocol and its SmPC.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 years;
* Clinical diagnosis of aTTP based on standard clinical and laboratory criteria (French Score ≥ 2): i.e., thrombotic microangiopathy syndrome with platelet count ≤ 30 G/L and serum creatinine ≤ 200 μmol/L; severe ADAMTS13 deficiency is not a requirement for inclusion of patients with a French score of 2 [31];
* Patient having read and understood the information letter and signed the Informed Consent Form. If the patient is unable to express his consent, the consent will be signed by his representative ((1) the trusted person, or failing that, (2) a family member, or (3) a close relative of the person concerned). In this case, consent to continue the study will subsequently be requested from the patient (article L1122-1-1 of the CSP);
* Patient affiliated with, or beneficiary of a social security (national health insurance) plan;
* For women:

  * Women of childbearing potential :

    * Effective contraception according to WHO definition (estrogen-progestin or intrauterine device or tubal ligation) since at least 1 month and;
    * Negative blood pregnancy test;
  * Women surgically sterile (absence of ovaries and/or uterus);
  * Postmenopausal women (non-medically induced amenorrhea for at least 12 months prior to the inclusion visit).

Exclusion Criteria:

* Platelet count > 100 G/L;
* Patients with a French score < 2 (a serum creatinine level > 200 μmol/L +/- associated with a platelet count > 30 G/L), in order to exclude possible cases of atypical hemolytic uremic syndrome;
* Known other causes of cytopenias and/or organ failure including but not limited to: uncontrolled cancer, chemotherapy, transplant, drugs, HIV at AIDS stage;
* Pregnant women (positive result from a blood pregnancy test) or patients with an imminent project of pregnancy; breastfeeding women (due to lack of pharmacological data for caplacizumab during pregnancy and breastfeeding);
* Congenital TTP;
* Clinically significant active bleeding or high risk of bleeding (excluding thrombocytopenia);
* Chronic treatment with anticoagulant that cannot be interrupted safely, including but not limited to: vitamin K antagonists, direct oral anticoagulant, low molecular weight heparin or heparin;
* Malignant hypertension;
* Contra-indication to CABLIVI 10 mg powder and solvent for solution for injection: hypersensitivity to caplacizumab or to any of the excipients;
* Contra-indication to PE treatment;
* Contra-indication to corticosteroid (= ((methyl)prednisone or (methyl)prednisolone)) or excipients;
* Contra-indication to rituximab or excipients and to its premedication;
* Person deprived of liberty by administrative or judicial decision or placed under judicial protection (guardianship or supervision);
* Participation in another drug interventional clinical trial within 30 days prior to inclusion and during the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the feasibility of a personalized caplacizumab regimen in aTTP based on ADAMTS13 activity monitoring assessed by a composite criteria including mortality, refractoriness and/or exacerbation at 30 days post-PE treatment | 30 days post-PE treatment
  composite endpoint defined by the occurrence of at least one the following events during the 30 days post-PE treatment: death, refractoriness or exacerbation.

SECONDARY OUTCOMES:
Response to treatment (platelet count recovery) | 30 days post-PE treatment
  to platelet count recovery (as defined by a platelet count ≥ 150 G/L with a subsequent interruption of daily PE within 5 days)
Durable remission achievement | 90 days post-PE treatment
  Occurrence of durable remission achievement (platelet count ≥ 150 G/L for ≥ 30 consecutive days following PE interruption);
Mortality at D90 post-PE treatment | 90 days post-PE treatment
  Occurrence of death within 90 days post-PE treatment
Refractoriness at D30 post-PE treatment | Day 30 post-PE treatment
  Occurrence of refractoriness at D30 post-PE treatment;
Exacerbation at D30 post-PE treatment | Day 30 post-PE treatment
  Occurrence of exacerbations at D30 post-PE treatment
Duration of plasma exchange (PE) treatment and the associated plasma volumes | 30 days
  Duration of daily PE with the corresponding plasma volume
Duration of plasma exchange (PE) treatment and the associated plasma | 30 days
  Total number of PE and the corresponding plasma volume during the full study drug treatment period
Occurrence of neurological sequelae treatment | Day 90 post-PE treatment
  Neurological assessment based on Rankin score
Evaluate the Quality of life | Day 90 post-PE treatment
  Quality of life based on global post-traumatic score (PCL-S SCALE) at baseline, D90 post-PE treatment
Evaluate the cost of the strategy | Day 90 post-PE treatment
  Costs of the patients' management (Direct hospital medical expenses, Suppléments, direct costs of home care, caplacizumab injections, rehospitalizations) of patients treated with the regimen according to the study
To perform a safety analysis | 90 days post-PE treatment
  Occurrence of AE and SAE during the study
Occurrence of cognitive sequelae treatment | Day 90 post-PE treatment
  Cognitive assessment based on MMS score

IPD SHARING:
Plan to Share IPD: No